CLINICAL TRIAL: NCT05028933
Title: Autologous T Cells Modified by Chimeric Antigen Receptor Targeting EpCAM for Clinical Research on Advanced Digestive System Malignancies
Brief Title: IMC001 for Clinical Research on Advanced Digestive System Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, professor, Zhejiang University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMC001-CT04
Record Dates: First submitted 2021-08-19; First posted 2021-08-31 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Advanced Hepatocellular Carcinoma; Advanced Colorectal Cancer; Advanced Gastric Cancer; Advanced Pancreatic Cancer
Keywords: EpCAM; CAR-T

STUDY DESIGN:
Intervention Model Description: single dose escalation The classic "3+3" dose escalation test. The starting dose refers to the results of the previous test of subsequent subjects. In this study, 3 increasing dose levels were set up, with 3 to 6 cases per dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EPCAM CAR-T (Experimental): The first stage: single dose escalation The classic "3+3" dose escalation test. The starting dose refers to the results of the previous test of subsequent subjects. In this study, 3 increasing dose levels were set up, with 3 to 6 cases per dose.
  * The first dose group is 3×10^5/kg, allowing 10% dose error.
  * The second dose group is 1×10^6/kg, allowing 10% dose error.
  * The third dose group is 3×10^6/kg, allowing 10% dose error. Each dose group must complete the DLT observation before entering the next dose group; when the first subject in the same dose group has no DLT observed for at least 14 days after cell infusion, the subsequent subjects can receive cell infusion.
  The second stage: combined radiofrequency/microwave ablation for the treatment of advanced digestive system malignant tumors with liver metastases
  Interventions: Drug: EPCAM CAR-T

INTERVENTIONS:
Drug: EPCAM CAR-T — Pretreatment with fludarabine and cyclophosphamide EpCAM CAR-T Cells infusion

SUMMARY:
A Phase I Clinical Study of Autologous T cells modified with chimeric antigen receptor targeting EpCAM ( EPCAM CAR-T) in Patients with malignant tumors of the digestive system (including advanced gastric cancer, colorectal cancer, liver cancer and pancreatic cancer) .

DETAILED DESCRIPTION:
This is a phase I open-label, single and multiple infusion, dose escalation/cohort expansion study to evaluate the safety, cell pharmacokinetics, and preliminary efficacy of EPCAM CAR-T, infused intravenously in subjects who have been diagnosed with advanced malignant tumors of the digestive system (including advanced gastric cancer, colorectal cancer, liver cancer and pancreatic cancer) and refractory or intolerant to current standard systemic treatment.

Primary objectives:

•To evaluate the safety and tolerability of EPCAM CAR-T infused intravenously at escalating doses in patients with advanced malignant tumors of the digestive system.

Secondary objectives:

1. The treatment of EpCAM CAR-T for patients with advanced digestive system malignancies, according to the dose-limiting toxicity and clinical response, including Possible side effects, determine the maximum tolerated dose (MTD), extended recommended dose (RDE) and/or recommended phase II dose (RP2D).
2. Assess the correlation between the pharmacodynamic (PD) biomarkers of IMC001 and clinical efficacy; EpCAM CAR-T expands and persists in vivo Correlation between sexual and pharmacodynamic (PD) biomarkers and adverse events.
3. To evaluate the preliminary anti-tumor efficacy of EpCAM CAR-T in patients with advanced digestive system malignancies. According to the evaluation criteria for the efficacy of solid tumors (RECIST) Version V.1.1, Evaluation Criteria for Efficacy of Immunotherapy for Solid Tumors (iRECIST), using objective response rate(ORR), duration of remission (DOR), disease control rate (DCR) and progression-free survival (PFS) description preliminary Anti-tumor activity.
4. The incidence of treatment-related adverse events.

Exploratory purpose:

1. Assess changes in immune status of EPCAM CAR-T treatment.
2. Assess the change of CTC in the peripheral blood of patients and the clearance effect of CAR-T cell treatment on CTC.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years old (including boundary value), both male and female.
2. The first stage requires patients with malignant tumors of the digestive system (including advanced gastric cancer, advanced colorectal cancer, advanced pancreatic cancer, advanced liver cancer) who have failed previous standard treatments and have no other feasible effective treatment methods. The documents for the diagnosis of advanced digestive system malignancies include imaging reports (CT/MRI) or pathological examination results. The second stage requires patients with liver metastases of advanced digestive system malignancies (including gastric cancer liver metastasis, colorectal cancer liver metastasis, and pancreatic cancer liver metastasis) who have previously failed standard treatment and have no other feasible effective treatment methods. The investigator can judge it. Perform radiofrequency/microwave ablation therapy. Documents for diagnosing liver metastases from advanced digestive system malignancies include imaging reports (CT/MRI) or pathological examination results.
3. The subject's expected survival period is ≥12 weeks.
4. According to the RECIST V.1.1 standard, subjects participating in the first phase of dose escalation must have at least one target lesion that can be evaluated stably. Participants participating in the second phase of EpCAM CAR-T infusion therapy combined with local radiofrequency/microwave ablation therapy must have at least one non-target disease in the liver that is suitable for radiofrequency/microwave ablation therapy.
5. The histological staining of EpCAM in the biopsy tumor tissue sample is positive.
6. Subjects in the second stage require Child-Pugh classification of liver function as A or B (score ≤ 7 points).
7. ECOG stamina score 0～1.
8. The subject has sufficient organ and bone marrow function. Laboratory screening must meet the following standards (refer to NCI CTCAE 5.0). All laboratory test results should be within the following stable range and there is no continuous supportive treatment.

   1. Blood test: white blood cell WBC≥1.5×10^9/L; platelet count PLT ≥60×10^9/L; hemoglobin content Hb ≥8.0g/dL; lymphocyte LYM≥0.4×10^9/L;
   2. Blood biochemistry: serum creatinine≤1.5×ULN, if serum creatinine>1.5×ULN, creatinine clearance rate>50mL/min (calculated according to Cockcroft-Gault formula); serum total bilirubin≤1.5×ULN, alanine Aminotransferase (ALT)≤2×ULN, aspartate aminotransferase (AST)≤2×ULN (ALT≤5×ULN in patients with liver metastasis or liver cancer, AST≤5×ULN).
   3. Amylase and lipase ≤ 1.5 × ULN;
   4. Routine urine examination: urine protein <2+
9. The left ventricular ejection fraction (LVEF)>45% in cardiac color Doppler ultrasound examination within one month.
10. Fertility status: female patients of childbearing age or male patients whose sexual partners are females of childbearing age are willing to take effective contraceptive measures from the signing of the informed consent form to 6 months after the last cell infusion (females of childbearing age include premenopausal women and premenopausal women). Women within 2 years after menopause).
11. The subject must sign and date a written informed consent form.
12. The subject must be willing and able to comply with the predetermined treatment plan, laboratory examination, follow-up and other research requirements.

Exclusion Criteria:

Subjects who meet any of the following conditions cannot be selected for this study;

1. Women during pregnancy and lactation.
2. Known history of human immunodeficiency virus (HIV) infection; acute or chronic active hepatitis B (HBsAg positive); acute or chronic active hepatitis C (HCV antibody positive). Syphilis antibody is positive; Epstein-Barr virus DNA quantitative> 500 copies; Cytomegalovirus (CMV) infection (IgM positive).
3. Severe infections that are active or poorly clinically controlled.
4. At present, there is a heart disease requiring treatment or a poorly controlled hypertension (defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure >90 mmHg after treatment with standardized antihypertensive drugs).
5. The presence of any of the following cardiac clinical symptoms or diseases:

   1. Unstable angina;
   2. Myocardial infarction occurred within 1 year;
   3. ECG at rest QTc>450ms (male) or QTc>470ms (female);
   4. The resting state ECG examination found abnormalities of important clinical significance (such as abnormal heart rate, conduction, morphological characteristics, etc.) or complete left bundle branch block or third-degree heart block or second-degree heart block or PR Interval> 250ms;
   5. There are factors that increase the risk of QTc prolongation and abnormal heart rate, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or sudden death of unexplained family members under 40 years old, or prolonged periods Period concomitant medication.
6. Abnormal blood coagulation function (INR>1.5×ULN), bleeding tendency or receiving thrombolysis or conventional anticoagulation therapy (such as warfarin or heparin), patients need long-term antiplatelet therapy (aspirin, dose> 300mg/day; Clopidogrel, dose>75mg/day).
7. Subjects who need to use corticosteroids or other immunosuppressive drugs for systemic therapy during the treatment period.
8. Before treatment, blood oxygen saturation ≤95% (referring to pulse oxygen detection).
9. Have received systemic steroids equivalent to >15 mg/day of prednisone within 2 weeks before apheresis, except for inhaled steroids.
10. Before the pretreatment of chemotherapy for removing lymphocytes, the subject developed a new arrhythmia, including but not limited to arrhythmia that cannot be controlled with drugs, hypotension that requires vasopressor, bacteria, fungi, or intravenous antibiotics that require intravenous antibiotics. Viral infection. Subjects who use test antibiotics to prevent infection are up to the investigator to determine whether participants can continue to participate in the test.
11. Known past or current hepatic encephalopathy requiring treatment; patients with current or history of central nervous system disease, such as epileptic seizures, cerebral ischemia/hemorrhage, dementia, cerebellar disease or any associated central nervous system involvement Autoimmune disease; central nervous system metastasis or meningeal metastasis with clinical symptoms, or other evidence that the patient's central nervous system metastasis or meningeal metastasis has not been controlled, and the investigator judged that it is not suitable for inclusion in the group.
12. The results of the imaging examination of the subjects in the second stage: the liver is replaced by tumors ≥50%, or the main portal vein tumor thrombus, or the tumor thrombus invades the mesenteric vein/inferior vena cava; or there are central or extensive non-metastatic lesions .
13. Patients who have had other malignant tumors before or at the same time, with the following exceptions:

    * Adequately treated basal cell or squamous cell carcinoma (enough wound healing is required before being enrolled in the study);
    * Cervical cancer or breast cancer in situ, after curative treatment, there is no sign of recurrence at least 3 years before the study;
    * The primary malignant tumor has been completely removed and completely remitted for ≥5 years.
14. Have received other CAR-T treatments and TCR-T treatments in the past.
15. Received anti-PD-1/PD-L1 monoclonal antibody treatment within 4 weeks before apheresis.
16. Subjects who have received other gene therapy in the past.
17. Subjects with severe mental disorders.
18. Participated in other clinical studies in the past month.
19. The researcher assesses that the subject is unable or unwilling to comply with the requirements of the research protocol.
20. The subject withdrew from the study due to various reasons and could not participate in the study again.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity （DLT） | 28 days
  Safety
Maximum Tolerated Dose（MTD） | 28 days
  Tolerability evaluation
Adverse Event(AE) | 28 days
  Incidence rate

SECONDARY OUTCOMES:
Number of Cells | 52 weeks
  Pharmacokinetics is the "Implantation endpoint" which is defined as the number of copies of the IMC001 DeoxyriboNucleic Acid（DNA）in peripheral blood detected at each visit after infusion until any two consecutive test results are negative or below the detection limit. Duration of IMC001 Cell persistence is the period from the day of infusion to the first negative test result or result lower than the detection limit
Treatment Emergent Adverse Events(TEAE) | Through study completion, an average of 3 years
  Incidence rate
Antitumor efficacy-objective response rate (ORR) | Through study completion, an average of 3 years
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause.
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause.
Antitumor efficacy-Progression-free survival (PFS) | Through study completion, an average of 3 years
  The period from the day when the subject receives the first study treatment to the first recorded tumor progression(whether treated or not) or death of any cause, which occurs first
Antitumor efficacy-Duration of response (DOR) | Through study completion, an average of 3 years
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause.
Antitumor efficacy-Overall survival (OS) | Through study completion, an average of 3 years
  The period from the first study treatment to any cause of death
Antitumor efficacy-Disease control rate (DCR) | Through study completion, an average of 3 years
  The number of cases in which response (PR + CR) and stable disease (SD) are achieved from the start of cell infusion/the total number of evaluable cases (%).
Number of circulating tumor cells (CTC) in peripheral blood | Through study completion, an average of 3 years
  The number of CTC before and after treatment was evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Weijia Fang, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (2):
- China (2):
  - Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - First affiliated hospital, School of Medicine, Zhejiang University, Hangzhou

IPD SHARING:
Plan to Share IPD: No